CLINICAL TRIAL: NCT00277784
Title: High-Resolution Ultrasound Imaging of the Retina and Choroid
Brief Title: High-Resolution Ultrasound Imaging of the Retina and Choroid for Detection on Age Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Ronald H. Silverman, PhD, Weill Cornell Medical College
Other Study IDs: AIUM #1-2005
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Age Related Macular Degeneration
Keywords: Age Related Macular Degeneration; Ultrasound; OCT; Eye
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Individuals with age related macular degeneration
  Interventions: Procedure: Ultrasound examination

INTERVENTIONS:
Procedure: Ultrasound examination — one ultrasound examination
  Other Names: High Frequency Ultrasound

SUMMARY:
The macula is the site of central vision within the retina. The retina is oxygenated by the underlying choroid. These tissues are less than 1 mm thick in total. While optical techniques can reveal much about the structure of the retina, ultrasound allows imaging of the choroid and deeper tissues. This study will investigate use of high frequency (20 MHz) ultrasound for imaging of the retina and choroid in patients with age-related macular degeneration, a prime cause of blindness. The investigation will involve use of novel post-processing methodologies to achieve maximum resolution of the fine tissue structures involved in this disease.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD), a condition affecting over 40% of individuals 70 years or age or more, causes progressive loss of central vision. Photocoagulation has long been used to slow the progress of AMD, but new vision-preserving methods are currently under investigation. Because destroyed photoreceptors are permanently lost, early management is essential for preservation of vision. The aim of this project will be to study AMD using a suite of new high-resolution ultrasound imaging techniques that have been developed. Specifically, high-resolution ultrasound will be used to generate images of the retina and choroid, including perfusion measurements using slow-flow methods developed by our research group. Ultrasound studies will be performed in conjunction with optical coherence tomography (OCT) imaging in a series of patients and age-matched control subjects with the aim of determining if choroidal thickness and/or perfusion might be used as an early indicator of AMD and thus aid in patient management.

We will study 20 subjects diagnosed with AMD. We will attempt to have an approximately equal number of subjects with wet and dry forms of AMD. A control group consisting of 20 non-AMD age-matched subjects will also be recruited. Ultrasound scan sequences will consist of B-mode images of the macula and surrounding tissues.

ELIGIBILITY:
Inclusion Criteria:

Age related macular degeneration age matched control

Exclusion Criteria:

none

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology practice
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Silverman, PhD, Principal Investigator — Weill Medical College of Cornell University; D. Jackson Coleman, MD, Study Chair — Weill Cornell Medical College - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Silverman RH. Ultrasound versus AC OCT. J Cataract Refract Surg. 2005 Aug;31(8):1475; author reply 1475-7. doi: 10.1016/j.jcrs.2005.08.011. No abstract available. PMID 16129261
- [Background] Coleman DJ, Silverman RH, Chabi A, Rondeau MJ, Shung KK, Cannata J, Lincoff H. High-resolution ultrasonic imaging of the posterior segment. Ophthalmology. 2004 Jul;111(7):1344-51. doi: 10.1016/j.ophtha.2003.10.029. PMID 15234135
- [Derived] Coleman DJ, Silverman RH, Rondeau MJ, Lloyd HO, Khanifar AA, Chan RV. Age-related macular degeneration: choroidal ischaemia? Br J Ophthalmol. 2013 Aug;97(8):1020-3. doi: 10.1136/bjophthalmol-2013-303143. Epub 2013 Jun 5. PMID 23740965